CLINICAL TRIAL: NCT04326166
Title: Multi-center, Open, Non-intervention and Observational Study to Evaluate the Efficacy and Safety of Suganon Tab. or Sugamet XR Tab. in Patients With Type 2 Diabetes
Brief Title: Observational Study to Evaluate the Efficacy and Safety of Suganon Tab. or Sugamet XR Tab.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DA1229_DM_OS
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one; Metformin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Patients who receive Double therapy or Insulin
  Interventions: Drug: Evogliptin
- Group B: Patients who receive DPP-4 inhibitor
  Interventions: Drug: Evogliptin
- Group C: Drug-naïve patients
  Interventions: Drug: Metformin and Evogliptin

INTERVENTIONS:
Drug: Evogliptin — Evogliptin
  Other Names: Suganon; Sugamet XR
  Groups: Group A
Drug: Evogliptin — Evogliptin
  Other Names: Suganon; Sugamet XR
  Groups: Group B
Drug: Metformin and Evogliptin — Metformin and Evogliptin
  Other Names: Suganon; Sugamet XR
  Groups: Group C

SUMMARY:
Multi-center, open, non-intervention and observational study to Evaluate the efficacy and safety of Suganon tab. or Sugamet XR tab. in patients with Type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

1. The subject is aged ≥19 years
2. The subject has type 2 diabetes mellitus

Exclusion Criteria:

1. The subject has a contraindication

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 DM patients
Sampling Method: Probability Sample
Enrollment: 1971 (Estimated)
Dates: Start 2020-03-25 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | at 12 weeks
  To assess change from baseline in HbA1c

SECONDARY OUTCOMES:
Change in HbA1c | at 24 weeks
  To assess change from baseline in HbA1c
The percentage of patients with HbA1c <7.0% and <6.5% | at 12 and 24 weeks
  To assess the percentage of patients with HbA1c <7.0% and <6.5%
Change in FPG | at 12 and 24 weeks
  To assess change from baseline in fasting plasma glucose (FPG)

CONTACTS AND LOCATIONS:
Locations (1):
- Sanggye paik pospital, Seoul, Nowon-gu, South Korea